CLINICAL TRIAL: NCT05538117
Title: Diagnostic Performance of Coronary Calcification Detection on CT Scan
Acronym: Calci-DT
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8697
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Thoracic pain; Acute coronary event; CT scan; Thoracic scan; Coronary calcifications; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
thoracic pain is one of the most frequent reasons for consulting the emergency room. Chest pain can be a sign of different pathologies with a wide range of severity, from life-threatening aortic dissection or myocardial infarction to chest pain during an anxiety attack. Efficient triage of patients is therefore a crucial issue for emergency physicians in order not to ignore an acute coronary event requiring early and specific management.

The investigators seek to evaluate whether a diagnostic strategy based on a thoracic CT scan to rule out coronary calcifications and a single troponin assay can exclude an acute coronary event with sufficient accuracy compared to usual management.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Patient admitted to the emergency room of the Nouvel Hôpital Civil in Strasbourg between 06/01/2021 and 12/31/2021 and presenting with typical chest pain <30min or atypical symptoms but non-eliminable cardiac origin.
* Patient with an initial assessment within the norms (ECG not modified, first troponin negative) and having performed a chest CT scan
* Patient who has not expressed his opposition to the reuse of his data for scientific research purposes.

Exclusion criteria:

- Patient who has expressed his opposition to the retrospective reuse of his data for scientific research purposes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) admitted to the emergency room of the Nouvel Hôpital Civil in Strasbourg between 06/01/2021 and 12/31/2021 and presenting with typical chest pain <30min or atypical symptoms but non-eliminable cardiac origin.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Ability of scan CT to detect coronary calcifications in patients presenting with thoracic pain to the emergency department | 30 minutes after onset of pain
  Presence on the scanner of calcifications 30 minutes after onset of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'accueil des urgences - CHU de Strasbourg - France, Strasbourg, France